CLINICAL TRIAL: NCT03824392
Title: A Randomized, Double-Blind, Placebo-Controlled Multiple Ascending Dose Study of Intravenous ATYR1923 in Patients With Pulmonary Sarcoidosis
Brief Title: Study of Intravenous ATYR1923 (Efzofitimod) for Pulmonary Sarcoidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Collaborators: Foundation for Sarcoidosis Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATYR1923-C-002
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Pulmonary Sarcoidosis; Resokine; Sarcoidosis; Granulomas; Inflammation; Lymphoproliferative Disorders; Interstitial Lung Disease; Neuropilin-2; Steroids; Oral corticosteroids; Immunomodulatory; tRNA Synthetase; ATYR1923 (efzofitimod)
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis; Granuloma; Inflammation; Lymphoproliferative Disorders; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: 36 participants with pulmonary sarcoidosis will be randomized into one of 3 sequential cohorts, each comprising 12 participants allocated 2:1 to efzofitimod:placebo matched to efzofitimod
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive placebo matched to efzofitimod via intravenous (IV) infusion every 4 weeks until Week 20.
  Interventions: Biological: Efzofitimod 1.0 mg/kg or Placebo; Biological: Efzofitimod 3.0 mg/kg or Placebo; Biological: Efzofitimod 5.0 mg/kg or Placebo
- Efzofitimod 1.0 mg/kg (Experimental): Participants will receive efzofitimod 1.0 milligrams/kilogram (mg/kg) via IV infusion every 4 weeks until Week 20.
  Interventions: Biological: Efzofitimod 1.0 mg/kg or Placebo
- Efzofitimod 3.0 mg/kg (Experimental): Participants will receive efzofitimod 3.0 mg/kg via IV infusion every 4 weeks until Week 20.
  Interventions: Biological: Efzofitimod 3.0 mg/kg or Placebo
- Efzofitimod 5.0 mg/kg (Experimental): Participants will receive efzofitimod 5.0 mg/kg via IV infusion every 4 weeks until Week 20.
  Interventions: Biological: Efzofitimod 5.0 mg/kg or Placebo

INTERVENTIONS:
Biological: Efzofitimod 1.0 mg/kg or Placebo — Participants to receive efzofitimod 1.0 mg/kg IV every 4 weeks or placebo matched to efzofitimod every 4 weeks
  Arms: Efzofitimod 1.0 mg/kg; Placebo
Biological: Efzofitimod 3.0 mg/kg or Placebo — Participants to receive efzofitimod 3.0 mg/kg IV every 4 weeks or placebo matched to efzofitimod every 4 weeks
  Arms: Efzofitimod 3.0 mg/kg; Placebo
Biological: Efzofitimod 5.0 mg/kg or Placebo — Participants to receive efzofitimod 5.0 mg/kg IV every 4 weeks or placebo matched to efzofitimod every 4 weeks
  Arms: Efzofitimod 5.0 mg/kg; Placebo

SUMMARY:
This randomized, double-blind, placebo matched to efzofitimod-controlled, study will evaluate the safety, tolerability, immunogenicity, pharmacokinetic (PK), and preliminary efficacy of multiple ascending doses of IV efzofitimod in participants with pulmonary sarcoidosis undergoing a protocol-guided oral corticosteroid (OCS) tapering regimen.This study will consist of 3 staggered multiple dose cohorts. Each eligible participant will participate in only one cohort during the study. Within each cohort, 12 participants will be randomized 2:1 to efzofitimod (N=8) or placebo matched to efzofitimod (N=4).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of pulmonary sarcoidosis for ≥6 months (cutaneous and ocular involvement allowed), defined as:

  * Histologically proven diagnosis of sarcoidosis by bronchoscopy, biopsy (any organ) or bronchioalveolar lavage
  * Parenchymal lung involvement by historical radiological evidence
* Must have symptomatic and/or active pulmonary sarcoidosis as evidenced by:

  * Modified Medical Research Council Dyspnea Scale grade of >= 1; and
  * Forced vital capacity ≥50%; and
* Receiving treatment with 10 to 25 mg/day of oral prednisone (or equivalent), at a stable dose for ≥4 weeks prior to Day 1, and capable of undergoing the protocol-specified steroid taper regimen.
* Body weight ≥45 kg and <160 kg.

Key Exclusion Criteria:

* Current disease presentation consistent with Lofgren's syndrome.
* History of severe allergic or anaphylactic reactions to therapeutic proteins or known sensitivity to efzofitimod or to its inactive components (L-histidine, sodium chloride, sucrose, L-methionine, and polysorbate-20).
* Treatment with biological immunomodulators such as tumor necrosis factor-alpha inhibitors.
* Current evidence of clinically significant cardiovascular, hepatic, renal, hematological, metabolic, or gastrointestinal disease, or has a condition that requires other treatment.
* Clinically significant pulmonary hypertension requiring vasodilator treatment.
* Any history of tuberculosis or evidence of active systemic non-tuberculosis fungal or mycobacterial infection within 1 year of Screening.
* History of clinically significant cardiac, neurological, gastrointestinal, and/or renal manifestations of sarcoidosis.
* Any condition that necessitated hospitalization within the 3 months prior to Day 1 or is likely to require so during the study.
* Participation in another clinical study of an investigational agent or device within 3 months (small molecules) / 6 months (biologics) or 5 half-lives (if known) of the agent, whichever is longer.
* History of or positive results of screening for hepatitis B, hepatitis C or human immunodeficiency virus.
* Is an active, heavy smoker of tobacco/nicotine-containing products (defined as >20 cigarettes/day or e-cigarette equivalent).
* Active substance abuse or history of substance abuse within the 12 months prior to Screening.
* Participant has received a live vaccination within 8 weeks before Day 1 or inoculation with a live vaccine is planned during study participation.
* Positive for Jo-1 antibodies (Ab) at Screening, or past history of Jo-1 Ab positivity.
* Significant and/or acute illness within 5 days prior to drug administration that may impact safety assessments, in the opinion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gennyne Walker, Study Director — aTyr Pharma, Inc.
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - aTyr Investigative Site, Northridge, California
  - National Jewish Health, Denver, Colorado
  - aTyr Investigative Site, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - aTyr Investigative Site, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Inova Fairfax Medical Center, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walker G, Adams R, Guy L, Chandrasekaran A, Kinnersley N, Ramesh P, Zhang L, Brown F, Niranjan V. Exposure-response analyses of efzofitimod in patients with pulmonary sarcoidosis. Front Pharmacol. 2023 Oct 3;14:1258236. doi: 10.3389/fphar.2023.1258236. eCollection 2023. PMID 37854715
- [Derived] Culver DA, Aryal S, Barney J, Hsia CCW, James WE, Maier LA, Marts LT, Obi ON, Sporn PHS, Sweiss NJ, Shukla S, Kinnersley N, Walker G, Baughman R. Efzofitimod for the Treatment of Pulmonary Sarcoidosis. Chest. 2023 Apr;163(4):881-890. doi: 10.1016/j.chest.2022.10.037. Epub 2022 Nov 8. PMID 36356657

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to efzofitimod via intravenous (IV) infusion every 4 weeks until Week 20.
- Efzofitimod 1.0 mg/kg: Participants received efzofitimod 1.0 milligrams/kilogram (mg/kg) via IV infusion every 4 weeks until Week 20.
- Efzofitimod 3.0 mg/kg: Participants received efzofitimod 3.0 mg/kg via IV infusion every 4 weeks until Week 20.
- Efzofitimod 5.0 mg/kg: Participants received efzofitimod 5.0 mg/kg via IV infusion every 4 weeks until Week 20.
Period: Overall Study
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
Started | 12 | 8 | 8 | 9
Received at Least 1 Dose of Study Drug | 12 | 8 | 8 | 9
Completed | 9 | 6 | 5 | 8
Not Completed | 3 | 2 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 1 | 0 | 0
Not completed — Participant Unable to Participate Due to COVID-19 Quarantine Restrictions | 2 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received any amount of study drug and were based on the actual treatment received, if this differs from that to which the participant was randomized.
Groups:
- Placebo: Participants received placebo matched to efzofitimod via IV infusion every 4 weeks until Week 20.
- Efzofitimod 1.0 mg/kg: Participants received efzofitimod 1.0 mg/kg via IV infusion every 4 weeks until Week 20.
- Total: Total of all reporting groups
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg | Total
Number analyzed (Participants) | 12 | 8 | 8 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.2) | 54.5 (11.3) | 51.8 (11.4) | 50.8 (9.2) | 52.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 4 | 5 | 20
  Male | 5 | 4 | 4 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 11 | 7 | 8 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 6 | 14
  White | 9 | 5 | 6 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs were defined as any adverse event or worsening of an existing condition after initiation of the investigational product and through 30 days after the participant's last study visit (study completion or early termination). SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
Number analyzed (Participants) | 12 | 8 | 8 | 9
Participants
  TEAEs | 10 | 8 | 7 | 8
  SAEs | 1 | 1 | 0 | 0

2. Secondary Outcome: Time-adjusted Area Under the Curve (AUC) of Background Oral Corticosteroid (OCS) Usage Over Study Period
Description: Time adjusted AUC is a measure of steroid burden and approximates the average daily OCS dose (mg/day) post-baseline for each participant. Time adjusted AUC was calculated by AUC divided by the number of days between first and last day of time interval of interest.
Time Frame: Baseline up to Week 24 (Day 1 to End of Dosing Period)
Population: The modified intent-to-treat (mITT) Set included all participants who had received any amount of study drug and were based on the randomized treatment, regardless of which treatment the participant actually received.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
Number analyzed (Participants) | 12 | 8 | 8 | 9
mg/day | 8.64 (4.20) | 6.83 (1.41) | 8.36 (3.68) | 7.43 (3.30)

3. Secondary Outcome: Number of Participants Who Achieved and Maintained The Targeted Tapered Dose of Prednisone 5 mg/Day (or Equivalent)
Time Frame: Baseline up to Week 24
Population: The mITT Set included all participants who had received any amount of study drug and were based on the randomized treatment, regardless of which treatment the participant actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
Number analyzed (Participants) | 12 | 8 | 8 | 9
Participants | 7 | 1 | 4 | 5

4. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (Anti-Efzofitimod)
Description: The number of all participants having drug reactive antibodies at any point in time (efzofitimod and placebo matched to efzofitimod) have been reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
Number analyzed (Participants) | 12 | 8 | 8 | 9
Participants | 1 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With at Least One Positive Anti-Jo-1 Antibodies Titers
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
Number analyzed (Participants) | 12 | 8 | 8 | 9
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: The Safety Set included all participants who received any amount of study drug and were based on the actual treatment received, if this differs from that to which the participant was randomized.
Arm/Group | Placebo | Efzofitimod 1.0 mg/kg | Efzofitimod 3.0 mg/kg | Efzofitimod 5.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 10/12 | 8/8 | 7/8 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Efzofitimod 1.0 mg/kg (N=8) | Efzofitimod 3.0 mg/kg (N=8) | Efzofitimod 5.0 mg/kg (N=9)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Efzofitimod 1.0 mg/kg (N=8) | Efzofitimod 3.0 mg/kg (N=8) | Efzofitimod 5.0 mg/kg (N=9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 4
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Vaccination site reaction (General disorders) | 0 | 0 | 0 | 1
Feeling jittery (General disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 2 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 1
Laboratory test abnormal (Investigations) | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Biopsy skin (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Narrow anterior chamber angle (Eye disorders) | 0 | 0 | 0 | 1
Scleritis (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03824392/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03824392/SAP_001.pdf